CLINICAL TRIAL: NCT00056446
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Study of Oxaliplatin/5-fluorouracil/Leucovorin With PTK787/ZK 222584 or Placebo in Patients With Previously Treated Metastatic Adenocarcinoma of the Colon or Rectum
Brief Title: Study of Oxaliplatin/5-FU/Leucovorin Plus Vatalanib Versus Oxaliplatin/5-FU/Leucovorin in Patients With Previously Treated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPTK787 0133/304946; NCT00068679 (obsolete NCT alias)
Record Dates: First submitted 2003-03-13; First posted 2003-03-14 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-01

CONDITIONS: Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms
Keywords: Colorectal Cancer; Oxaliplatin; VEGF inhibitor; Vatalanib; PTK787; Colon Cancer; Colorectal Carcinoma; Rectal Cancer; Colorectal Tumor
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oxaliplatin/5-FU/LV and PTK787/ZK 222584
  Interventions: Drug: Vatalanib
- 2 (Placebo Comparator): Oxaliplatin/5-FU/LV and placebo
  Interventions: Drug: Vatalanib

INTERVENTIONS:
Drug: Vatalanib
  Other Names: PTK787/ZK 222584

SUMMARY:
The purpose of this study is to compare treatment with oxaliplatin/5-FU/leucovorin plus vatalanib versus oxaliplatin/5-FU/leucovorin plus placebo in patients with colorectal cancer that has spread to other organs and whose disease has worsened after treatment with irinotecan.

ELIGIBILITY:
Inclusion criteria

* Confirmed adenocarcinoma of the colon or rectum in patients with metastatic disease
* One prior chemotherapy regimen with irinotecan and 5FU
* Evidence of progressive disease within 6 months after last dose of irinotecan
* WHO Performance Status of 0, 1, or 2
* Measurable tumors
* Adequate hematologic status, liver and kidney function
* Life expectancy greater than 12 weeks
* Written informed consent obtained

Exclusion criteria

* History or presence of central nervous system disease
* Patients with a history of another primary cancer within 5 years
* Prior chemotherapy within 3 weeks before entry to study
* Major surgery within 4 weeks or minor surgery within 2 weeks before entry to study
* Investigational drugs within 4 weeks before entry to study
* Prior therapy with oxaliplatin
* Peripheral neuropathy with functional impairment
* Female patients who are pregnant or breast feeding
* Any severe or uncontrolled medical condition which could prevent participation in study
* Chronic kidney disease
* Acute or chronic liver disease
* Patients taking Coumadin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 2003-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | throughout duration of study

SECONDARY OUTCOMES:
Progression free survival | throughout duration of study
Time to progression | throughout duration of study
Time to treatment failure | throughout duration of study
Tumor response rate | throughout duration of study
Tolerability and safety profile | throughout duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis/Schering AG, Germany, Study Chair — Novartis / Schering AG Germany
Locations (239):
- United States (143):
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Arizona Clinical Research Center, Tucson, Arizona
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Arkansas Cancer Research Center, Little Rock, Arkansas
  - Little Rock Hematology & Oncology, Little Rock, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Providence St. Joseph Medical Center, Burbank, California
  - Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - California Oncology of the Central Valley, Fresno, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - Glendale Adventist Medical Center, Glendale, California
  - Scripps Green Hospital, La Jolla, California
  - Wilshire Oncology Medical Group, La Verne, California
  - Pacific Shores Medical Group, Long Beach, California
  - USC Norris Cancer Center, Los Angeles, California
  - Synergy Hematology-Oncology Medical Associates, Los Angeles, California
  - Novartis Investigative Site, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - Eddie Hong-Lung Hu, M.D., Monterey Park, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Medical Oncology Care Associates, Orange, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Sierra View District Hospital, Porterville, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Sansum Santa Barbara Foundation Medical Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - San Diego Cancer Center Medical Group, Vista, California
  - Mile High Oncology, Denver, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Manchester Hematology/Oncology Assoc., Manchester, Connecticut
  - Washington Oncology/Hematology Center, Washington D.C., District of Columbia
  - The Center for Hematology and Oncology, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Hematology Oncology Associates, Lake Worth, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Oncology/Hematology Group of South Florida, Miami, Florida
  - Hematology Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Florida Medical Clinic, Zephyrhills, Florida
  - Atlanta Cancer Care, Marietta, Georgia
  - Office of Research, Savannah, Georgia
  - Coastal Hematology & Oncology, Savannah, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - University of Chicago medical Center, Hematology/Oncology, Chicago, Illinois
  - Oncology Hematology Associates of Central Illinois, PC, Peoria, Illinois
  - Northshore Cancer Research Association, Skokie, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Fort Wayne Medical Oncology & Hematology, Inc., Fort Wayne, Indiana
  - Munster Community Hospital, Munster, Indiana
  - Cotton O'Neil Oncology Clinic, Topeka, Kansas
  - Vijay Raghaven, M.D., Louisville, Kentucky
  - Owensboro Medical Health System, Owensboro, Kentucky
  - Cabrini Center for Cancer Care, Alexandria, Louisiana
  - LSU Medical Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Maine Center for Cancer Medicine & Blood Disorders, Scarborough, Maine
  - St. Agnes Healthcare, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Kaiser Permanente, Rockville, Maryland
  - Fallon Clinic at Worcester Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health -- Cook Research Dept., Grand Rapids, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Providence Cancer Center, Southfield, Michigan
  - Minnesota CGOP, Minneapolis, Minnesota
  - Heartland Hematology, Kansas City, Missouri
  - Missouri Cancer Care, PC, Saint Charles, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services Incorporated, St Louis, Missouri
  - North Central Montana Professional Building, Great Falls, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Center, Las Vegas, Nevada
  - NH Oncology-Hematology, PA, Hooksett, New Hampshire
  - Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - St. Barnabas Cancer Center, Livingston, New Jersey
  - Hematology Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - Cooper Cancer Center, Voorhees Township, New Jersey
  - Hematology/Oncology Associates, Albuquerque, New Mexico
  - New Mexico Oncology/Hematology, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology/Oncology Associates of Central NY, East Syracuse, New York
  - Queens Medical Associates, PC, Fresh Meadows, New York
  - Charles R. Wood Cancer Center, Glens Falls, New York
  - North Shore University Hospital, Manhasset, New York
  - St. Vincent's Catholic Medical Centers of New York, New York, New York
  - Hematology-Oncology Associates of Rockland, Nyack, New York
  - Pluta Cancer Center, Rochester, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Hematology/Oncology Associates, Charlotte, North Carolina
  - Nashat Gabrail, M.D., Canton, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus CCOP, Columbus, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Oncology, Inc., Tulsa, Oklahoma
  - Consultants in Medical Oncology & Hematology, Drexel Hill, Pennsylvania
  - Hematology & Oncology Associates of NE PA, Dunmore, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Monongahela Valley Hospital, Monongahela, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Pavillion, Pittsburgh, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - South Carolina Oncology Associates, Columbia, South Carolina
  - WJB Dom VAMC, Columbia, South Carolina
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Clarksville Regional Hematology/Oncology, Clarksville, Tennessee
  - The Jones Clinic, Germantown, Tennessee
  - Baptist Regional Cancer Center, Knoxville, Tennessee
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Center for Oncology Research & Treatment, Dallas, Texas
  - Clinical Hematology & Oncology, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - H. Alejandro Preti, M.D., PA, Houston, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - South Texas Oncology & Hematology, San Antonio, Texas
  - Scott & White Hospital, Temple, Texas
  - Northern Utah Cancer Associates, Ogden, Utah
  - Southwestern Vermont Health Care, Bennington, Vermont
  - Virginia Oncology Associates, Norfolk, Virginia
  - Cancer Treatment Centers of America in Hampton Roads, Portsmouth, Virginia
  - Western Washington Clinic, Everett, Washington
  - Cascade Cancer Center, Kirkland, Washington
  - Rainier Oncology, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - West Virginia University Health Sciences Center, Morgantown, West Virginia
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Kettle Morain Oncology, West Bend, Wisconsin
- Australia (2):
  - Novartis Investigative Site, Frankston
  - Novartis Investigative Site, Woodville South
- Novartis Investigative Site, Sankt Veit an der Glan, Austria
- Belgium (6):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Wilrijk
- Brazil (4):
  - Novartis Investigative Site, Porto Alegre RS
  - Novartis Investigative Site, Salvador - Ba
  - Novartis Investigative Site, Salvador, Bahia
  - Novartis Investigative Site, São Paulo
- Canada (18):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Penticton, British Columbia
  - Novartis Investigative Site, Winnepeg, Manitoba
  - Novartis Investigative Site, Sydney, Nova Scotia
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Sainte-Foy, Ontario
  - Novartis Investigative Site, St. Catharines, Ontario
  - Novartis Investigative Site, Thunder Bay, Ontario
  - Toronto, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- France (10):
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Boulogne
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (17):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wiesbaden
- Novartis Investigative Site, Chai Wan, Hong Kong
- Italy (10):
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Bergamo
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Cremona
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Livorno
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Reggio Emilia
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Rozzano
- New Zealand (3):
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, Wellington
- Portugal (2):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
- Novartis Investigative Site, Bratislava, Slovakia
- Spain (5):
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Elche
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Zaragoza
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Thun
- Taiwan (7):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Keelung
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (5):
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

REFERENCES:
- [Result] Van Cutsem E, Bajetta E, Valle J, Kohne CH, Hecht JR, Moore M, Germond C, Berg W, Chen BL, Jalava T, Lebwohl D, Meinhardt G, Laurent D, Lin E. Randomized, placebo-controlled, phase III study of oxaliplatin, fluorouracil, and leucovorin with or without PTK787/ZK 222584 in patients with previously treated metastatic colorectal adenocarcinoma. J Clin Oncol. 2011 May 20;29(15):2004-10. doi: 10.1200/JCO.2010.29.5436. Epub 2011 Apr 4. PMID 21464401